| Statistical Analy | vsis Plan | J2G-MC-J | JZJU V | Version | 1.0 |
|-------------------|-----------|----------|--------|---------|-----|
|-------------------|-----------|----------|--------|---------|-----|

An Open-Label, Randomized Study to Evaluate the Relative Bioavailbility of Selpercatinib in 3 Formulations for Pediatric Use

NCT05136404

Approval Date: 09-Nov-2021

# STATISTICAL ANALYSIS PLAN

# An Open-Label, Randomized Study to Evaluate the Relative Bioavailability of Selpercatinib in 3 Formulations for Pediatric Use

Statistical Analysis Plan Status: Final Statistical Analysis Plan Version: 1.0 Statistical Analysis Plan Date: 04 November 2021

Investigational Medicinal Product: LY3527723

Protocol Reference: J2G-MC-JZJU Labcorp Study: 8445329

Clinical Phase I

Approval Date: 09-Nov-2021 GMT

# 1. TABLE OF CONTENTS

| 1. | TABLE ( | OF CONTENTS | 2 |
|---|---|---|---|
| 2. | ABBREV | /IATIONS | 3 |
| 3. | INTROD | UCTION | 5 |
| 4. | STUDY | OBJECTIVES AND ENDPOINTS | 5 |
| <b>5.</b> | STUDY | DESIGN | 6 |
| | 5.1 Scree | ening | 6 |
| | 5.2 Trea | tment and Assessment Period | 6 |
| 6. | | MENTS | |
| <b>7.</b> | SAMPLE | E SIZE JUSTIFICATION | 7 |
| 8. | DEFINIT | TION OF ANALYSIS POPULATIONS | 7 |
| 9. | STATIST | TICAL METHODOLOGY | 8 |
| | 9.1 Gene | eral | 8 |
| | | ographics and Participant Disposition | |
| | 9.3 Phar | macokinetic Assessment | 8 |
| | 9.3.1 | Pharmacokinetic Analysis. | 8 |
| | 9.3.2 | Pharmacokinetic Statistical Methodology | . 12 |
| | 9.4 Safet | ry and Tolerability Assessments | |
| | 9.4.1 | Adverse events | . 13 |
| | 9.4.2 | Concomitant medication. | . 13 |
| | 9.4.3 | Clinical laboratory parameters | . 13 |
| | 9.4.4 | Vital signs | |
| | 9.4.5 | Electrocardiogram (ECG). | . 13 |
| | 9.4.6 | Hepatic Monitoring | . 14 |
| | 9.4.7 | Palatability Questionnaires | . 14 |
| | 9.4.8 | Other assessments | . 14 |
| | 9.4.9 | Safety and Tolerability Statistical Methodology | . 14 |
| | | M ANALYSES | . 14 |
| | | ES FROM THE PROTOCOL SPECIFIED STATISTICAL ANALYSES | |
| | | NCES | |
| 13. | | RESENTATION | |
| | | ved Parameters | |
| | | ing Data | |
| | 13.3 Insufficient Data for Presentation | | |
| 14. | | DICES | |
| | Appendix | 1: Document History | . 16 |

Statistical Analysis Plan CONFIDENTIAL Labcorp Study: 8445329 Protocol Reference: J2G-MC-JZJU

# 2. ABBREVIATIONS

Abbreviations pertain to the Statistical Analysis Plan (SAP) only (not the tables, figures and listings [TFLs]).

AE Adverse event

AUC Area under the concentration versus time curve

 $AUC(0-\infty)$  Area under the concentration versus time curve from time zero to

infinity

AUC(0-t<sub>last</sub>) Area under the concentration versus time curve from time zero to

time t, where t is the last time point with a measurable concentration

BQL Below the lower limit of quantitation

CI Confidence interval

CL/F Apparent total body clearance of drug calculated after extra-vascular

administration

C<sub>last</sub> Last predicted observed drug concentration

C<sub>max</sub> Maximum observed drug concentration

CRU Clinical Research Unit
CSR Clinical Study Report
CV% Coefficient of variation

ECG Electrocardiogram

ICH International Conference on Harmonisation

MedDRA Medical Dictionary for Regulatory Activities

PFOS Powder for oral suspension

PK Pharmacokinetic

RTU Ready to use

SAE Serious adverse event
SAP Statistical Analysis Plan

SD Standard deviation

 $t_{1/2}$  Half-life associated with the terminal rate constant ( $\lambda_z$ ) in non-

compartmental analysis

TEAE Treatment-emergent adverse event

TFLs Tables, Figures, and Listings

t<sub>max</sub> Time of maximum observed drug concentration

| V <sub>ss</sub> /F | Apparent volume of distribution at steady state after extravascular administration |
|---|---|
| V <sub>z</sub> /F | Apparent volume of distribution during the terminal phase after extra-vascular administration |
| WHO | World Health Organization |

CONFIDENTIAL

Protocol Reference: J2G-MC-JZJU

# 3. INTRODUCTION

This SAP has been developed after review of the Clinical Study Protocol (final version dated 19 July 2021), and protocol amendment (a) (final version dated 07 September 2021).

This SAP describes the planned analysis of the safety, tolerability and pharmacokinetic (PK) data from this study. A detailed description of the planned TFLs to be presented in the clinical study report (CSR) is provided in the accompanying TFL shell document.

The intent of this document is to provide guidance for the statistical and PK analyses of data. In general, the analyses are based on information from the protocol, unless they have been modified by agreement with Eli Lilly and Company. A limited amount of information concerning this study (e.g., objectives, study design) is given to help the reader's interpretation. For open-label studies, this SAP must be signed off prior to first participant visit for this study. When the SAP and TFL shells are agreed upon and finalized, they will serve as the template for this study's CSR.

This SAP supersedes the statistical considerations identified in the protocol; where considerations are substantially different, they will be so identified. If additional analyses are required to supplement the planned analyses described in this SAP, they may be performed and will be identified in the CSR. Any substantial deviations from this SAP will be agreed upon with Eli Lilly and Company and identified in the CSR. Any minor deviations from the TFLs may not be documented in the CSR.

This SAP is written with consideration of the recommendations outlined in the International Conference on Harmonisation (ICH) E9 Guideline entitled Guidance for Industry: Statistical Principles for Clinical Trials<sup>1</sup> and the ICH E3 Guideline entitled Guidance for Industry: Structure and Content of Clinical Study Reports<sup>2</sup>.

# 4. STUDY OBJECTIVES AND ENDPOINTS

| Objectives | Endpoints |
|---|---|
| Primary | |
| To evaluate the relative bioavailability of<br>RTU (ready to use) and PFOS (powder for<br>oral suspension) suspensions compared to<br>the capsule formulation | <ul> <li>Maximum observed drug concentration<br/>(C<sub>max</sub>), area under the concentration<br/>versus time curve from time zero to<br/>infinity (AUC[0-∞]), area from under the<br/>concertation versus time curve from time<br/>zero to time t (AUC0-t<sub>last</sub>), and time to<br/>maximum observed drug concentration<br/>(t<sub>max</sub>) of selpercatinib</li> </ul> |
| Secondary | |
| To evaluate the safety and tolerability of a single 20-mg oral dose of selpercatinib RTU and PFOS suspensions | Summary of the number, severity, and type of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) |

| • [ | To assess the palatability of selpercatinib | • | Responses to palatability questionnaire |
|---|---|---|---|
| ] | RTU and PFOS suspensions | | (RTU suspension only) |

# 5. STUDY DESIGN

Study J2G-MC-JZJU (JZJU) will be an open-label, Phase 1 randomized, 3-formulation, 3-period, crossover study in adult heathy male and female participants. The RTU 20-mg suspension and the PFOS 20 mg/mL formulation will be compared to the 20 mg capsule formulation.

Figure 1 below illustrates the study design.



Figure 1: J2G-MC-JZJU Study Schema

Safety assessments, including adverse events (AEs), concomitant medications, medical assessments, clinical laboratory tests, vital signs, and electrocardiograms (ECGs), and blood sampling for PK, will be performed.

### 5.1 **Screening**

All participants will be screened within 28 days prior to enrolment.

### 5.2 **Treatment and Assessment Period**

Participants will be admitted to the clinical research unit (CRU) on Day -1. On the morning of Day 1, participants will be randomized to 1 of 3 treatment sequences and will receive single doses of 20 mg selpercatinib on each of Days 1, 8, and 15 as either the RTU suspension, the PFOS, or the capsule, and will be dosed according to the randomization sequence following an overnight fast of at least 10 hours.

The treatment sequences to be used are shown in Figure 2:



Figure 2: Treatment Sequences for Study J2G-MC-JZJU

There will be a washout of 7 days between doses of selpercatinib. Participants will remain resident at the CRU for the full duration of the treatment period (i.e., up to Day 21).

# 6. TREATMENTS

The following is a list of the study treatment abbreviations that will be used in the TFLs.

| Study Treatment Name | Abbreviation | Treatment order in TFL |
|------------------------------------|--------------|------------------------|
| 20 mg selpercatinib capsule | Capsule | 1 |
| RTU selpercatinib 20 mg Suspension | RTU | 2 |
| 20 mg/mL selpercatinib PFOS | PFOS | 3 |

PFOS = powder for oral suspension, RTU = ready to use

# 7. SAMPLE SIZE JUSTIFICATION

Up to approximately 42 participants will be enrolled to ensure that at least approximately 36 participants complete the study. The sample size for this study is justified based on a precision for the ratio of geometric means and it is represented by the half-width of the 90% confidence interval (CI) of the point estimate on the logarithmic scale. Based on an intra-participant variability of 70% (LOXO-RET-19075), with a probability of 90%, a 90% CI for the ratio of the geometric means for C<sub>max</sub> and area under the concentration versus time curve (AUC) will be obtained with a precision about 0.288 in the log scale, which corresponds to approximately 0.334 in the natural scale.

# 8. DEFINITION OF ANALYSIS POPULATIONS

The "Safety" population will consist of all enrolled participants who received at least one dose of selpercatinib, whether or not they completed all protocol requirement.

The "Pharmacokinetic" population will consist of all participants who received at least one dose of selpercatinib and have evaluable PK data. Participants may be excluded from the PK summary statistics and statistical analysis if a participant has an AE of vomiting that occurs at or before 2 times median  $t_{max}$ .

CONFIDENTIAL Protocol Reference: J2G-MC-JZJU

All protocol deviations that occur during the study will be considered for their severity/impact and will be taken into consideration when participants are assigned to analysis populations.

# 9. STATISTICAL METHODOLOGY

### 9.1 General

Data listings will be provided for all data that is databased. Summary statistics and statistical analysis will only be presented for data where detailed in this SAP. For continuous data, summary statistics will include the arithmetic mean, arithmetic standard deviation (SD), median, minimum, maximum and n (number of subjects); for log-normal data (e.g. the PK parameters: AUCs and C<sub>max</sub>) the geometric mean and geometric coefficient of variation (CV%) will also be presented. For categorical data, frequency count and percentages will be presented. Data listings will be provided for all participants up to the point of withdrawal, with any participants excluded from the relevant population highlighted. Summary statistics and statistical analyses will generally only be performed for participants included in the relevant analysis population. For the calculation of summary statistics and statistical analysis, unrounded data will be used.

Mean change from baseline is the mean of all individual participants' change from baseline values. Each individual change from baseline will be calculated by subtracting the individual participant's baseline value from the value at the timepoint. The individual participant's change from baseline values will be used to calculate the mean change from baseline using a SAS procedure such as Proc Univariate.

Data analysis will be performed using SAS® Version 9.4 or greater.

### 9.2 **Demographics and Participant Disposition**

Participant disposition will be summarized and listed. The demographic variables age, sex, race, ethnicity, country of enrolment, site ID, body weight, height and body mass index will be summarized and listed. All other demographic variables will be listed only.

### 9.3 **Pharmacokinetic Assessment**

### Pharmacokinetic Analysis 9.3.1

Noncompartmental methods applied with a validated software program (Phoenix WinNonlin Version 8.1 or later) to the plasma concentrations of selpercatinib will be used to determine the following PK parameters, when possible:

| Parameter | Units | Definition area under the concentration versus time curve from time zero to time t, where t is the last time point with a measurable concentration |
|---|---|---|
| AUC(0-t <sub>last</sub> ) | ng.h/mL | |
| $AUC(0-\infty)$ | ng.h/mL | area under the concentration versus time curve from time zero to infinity |
| $C_{max}$ | ng/mL | maximum observed drug concentration |
| $t_{max}$ | h | time of maximum observed drug concentration |
| $t_{1/2}$ | h | half-life associated with the terminal rate constant $(\lambda_z)$ in non-compartmental analysis |
| CL/F | L/h | apparent total body clearance of drug calculated after extra-vascular administration |
| V <sub>Z</sub> /F | L | apparent volume of distribution during the terminal phase after extra-vascular administration |
| V <sub>SS</sub> /F | L | apparent volume of distribution at steady state after extra-vascular administration |

Additional PK parameters may be calculated, as appropriate.

The software and version used for the final analyses will be specified in the CSR. Any exceptions or special handling of data will be clearly documented within the final CSR.

Formatting of tables, figures and abbreviations will follow the Eli Lilly Global PK/PD/TS Tool: NON-COMPARTMENTAL PHARMACOKINETIC STYLE GUIDE. The version of the tool effective at the time of PK analysis will be followed.

# **General PK Parameter Rules**

- Actual sampling times will be used in the final analyses of individual PK parameters, except for non-bolus pre-dose sampling times which will be set to zero.
- $C_{max}$  and  $t_{max}$  will be reported from observed values. If  $C_{max}$  occurs at more than one time point, t<sub>max</sub> will be assigned to the first occurrence of C<sub>max</sub>.
- AUC parameters will be calculated using a combination of the linear and logarithmic trapezoidal methods (linear-log trapezoidal rule). The linear trapezoidal method will be applied up to  $t_{max}$  and then the logarithmic trapezoidal method will be used after  $t_{max}$ . The minimum requirement for the calculation of AUC will be the inclusion of at least three consecutive plasma concentrations above the lower limit of quantification, with at least one of these concentrations following  $C_{max}$ .
- The  $t_{1/2}$  will be calculated, when appropriate, based on the apparent terminal log-linear portion of the concentration-time curve. The start of the terminal elimination phase for each subject will be defined by visual inspection and generally will be the first point at which there is no systematic deviation from the log-linear decline in plasma concentrations. Half-life will only be calculated when a reliable estimate for this

parameter can be obtained comprising of at least 3 data points. If  $t_{1/2}$  is estimated over a time window of less than 2 half-lives, the values will be flagged in the data listings. Any  $t_{1/2}$  value excluded from summary statistics will be documented in the footnote of the summary table.

- A uniform weighting scheme will be used in the regression analysis of the terminal loglinear portion of the concentration-time curve.
- The parameters based on last predicted observed drug concentration (C<sub>last</sub>) will be reported (except in bioequivalence and bioavailability studies, where only the observed parameters will be reported).

# **Individual PK Parameter Rules**

- Only quantifiable concentrations will be used to calculate PK Parameters with the exception of special handling of certain concentrations reported below the lower limit of quantitation (BQL). Plasma concentrations reported as BQL will be set to a value of zero when all of the following conditions are met:
  - The compound is non-endogenous.
  - The samples are from the initial dose period for a subject or from a subsequent dose period following a suitable wash-out period.
  - o The time points occur before the first quantifiable concentration.
- All other BQL concentrations that do not meet the above criteria will be set to missing.
- Also, where two or more consecutive concentrations are BQL towards the end of a profile, the profile will be deemed to have terminated and therefore any further quantifiable concentrations will be set to missing for the calculation of the PK parameters unless it is considered to be a true characteristic of the profile of the drug.

# **Individual Concentration vs. Time Profiles**

- Individual concentrations will be plotted utilizing actual sampling times.
- The terminal point selections will be indicated on a semi-logarithmic plot.

# **Average Concentration vs. Time Profiles**

- The average concentration profiles will be graphed using scheduled (nominal) sampling times.
- The average concentration profiles will be graphed using arithmetic average concentrations.

- The pre-dose average concentration for single-dose data from non-endogenous compounds will be set to zero. Otherwise, only quantifiable concentrations will be used to calculate average concentrations.
- Concentrations at a sampling time exceeding the sampling time window specified in the protocol, or  $\pm$  10%, will be excluded from the average concentration profiles.
- Concentrations excluded from the mean calculation will be documented in the final CSR.
- A concentration average will be plotted for a given sampling time only if 2/3 of the individual data at the time point have quantifiable measurements that are within the sampling time window specified in the protocol or  $\pm$  10%. An average concentration estimated with less than 2/3 but more than 3 data points may be displayed on the mean concentration plot if determined to be appropriate and will be documented within the final CSR.

# **Treatment of Outliers during Pharmacokinetic Analysis**

Application of this procedure to all PK analyses is not a requirement. Rather, this procedure provides justification for exclusion of data when scientifically appropriate. This procedure describes the methodology for identifying an individual value as an outlier for potential exclusion, but does not require that the value be excluded from analysis. The following methodology will not be used to exclude complete profiles from analysis.

# Data within an Individual Profile

A value within an individual profile may be excluded from analysis if any of the following criteria are met:

- For PK profiles during multiple dosing, the concentration of the pre-dose sample exceeds all measured concentrations for that individual in the subsequent post-dose samples.
- For PK profiles during single dosing of non-endogenous compounds, the concentration in a pre-dose sample is quantifiable.
- For any questionable datum that does not satisfy the above criteria, the profile will be evaluated and results reported with and without the suspected datum.

# Data between Individual Profiles

- 1. If n<6, then the dataset is too small to conduct a reliable range test. Data will be analyzed with and without the atypical value, and both sets of results will be reported.
- 2. If n≥6, then an objective outlier test will be used to compare the atypical value to other values included in that calculation:
  - a. Transform all values in the calculation to the logarithmic domain.

- b. Find the most extreme value from the arithmetic mean of the log transformed values and exclude that value from the dataset.
- c. Calculate the lower and upper bounds of the range defined by the arithmetic mean  $\pm 3*SD$  of the remaining log-transformed values.
- d. If the extreme value is within the range of arithmetic mean  $\pm 3*SD$ , then it is not an outlier and will be retained in the dataset.
- e. If the extreme value is outside the range of arithmetic mean  $\pm 3*SD$ , then it is an outlier and will be excluded from analysis.

If the remaining dataset contains another atypical datum suspected to be an outlier and  $n \ge 6$  following the exclusion, then repeat step 2 above. This evaluation may be repeated as many times as necessary, excluding only one suspected outlier in each iteration, until all data remaining in the dataset fall within the range of arithmetic mean  $\pm 3*SD$  of the log-transformed values.

# Reporting of Excluded Values

Individual values excluded as outliers will be documented in the final CSR. Approval of the final CSR will connote approval of the exclusion.

# 9.3.2 Pharmacokinetic Statistical Methodology

PK parameters will be evaluated to estimate relative bioavailability of the RTU and PFOS suspensions compared to the capsule formulation.

Log-transformed  $C_{max}$ ,  $AUC(0-\infty)$ , and  $AUC(0-t_{last})$  parameters will be evaluated in a linear mixed effect model with fixed effects for treatment formulation, period, sequence, and a random effect for participant. The treatment differences between RTU (test) and PFOS (test), and the capsule (reference) formulations will be back-transformed to present the ratios of geometric least squares means and the corresponding 90% CIs.



The  $t_{max}$  will be analyzed using a Wilcoxon signed rank test. Estimates of the median difference based on the individual paired differences, 90% CIs, and p-values from the Wilcoxon test will be calculated.

### 9.4 Safety and Tolerability Assessments

### 9.4.1 **Adverse events**

Where changes in severity are recorded in the CRF, each separate severity of the AE will be reported in the listings, only the most severe will be used in the summary tables. A pre-existing condition is defined as a condition that starts before the participant has provided written informed consent and is ongoing at consent. A non-treatment emergent AE is defined as an AE which starts after informed consent but prior to dosing. A TEAE is defined as an AE which occurs postdose or which is present prior to dosing and becomes more severe postdose.

All AEs will be listed. TEAEs will be summarized by treatment, severity and relationship to the study drug. The frequency (the number of AEs, the number of participants experiencing an AE and the percentage of participants experiencing an AE) of TEAEs will be summarized by treatment, Medical Dictionary for Regulatory Activities (MedDRA) version 24.0 system organ class and preferred term. The summary and frequency AE tables will be presented for all causalities and those considered related to the study drug by the investigator. Any SAEs will be listed.

Discontinuations due to AEs will be listed.

### **Concomitant medication** 9.4.2

Concomitant medication will be coded using the WHO drug dictionary (Version March 2021). Concomitant medication will be listed.

### 9.4.3 Clinical laboratory parameters

All clinical chemistry and hematology data will be summarized by parameter and treatment, and listed. Urinalysis data will be listed. Additionally, clinical chemistry, hematology and urinalysis data outside the reference ranges will be listed and flagged on individual participant data listings.

### 9.4.4 Vital signs

Vital signs data will be summarized by treatment together with changes from baseline, where baseline is defined as the Day 1, Day 8, or Day 15 predose (as appropriate) assessment. Figures of mean vital signs and mean changes from baseline profiles will be presented by treatment, for 0 (predose) to 96 h (Day 5/11/19) postdose.

Values for individual participants will be listed.

### 9.4.5 Electrocardiogram (ECG)

ECGs will be performed for safety monitoring purposes only and will not be presented. Any clinically significant findings from ECGs will be reported as an AE.

# 9.4.6 Hepatic Monitoring

If a participant experiences elevated laboratory parameters, as detailed in Section 8.2.6.1 of the protocol, additional tests will be performed to confirm the abnormality. Additional safety data may be collected if required, as defined in the protocol. Where applicable, the following will be presented.

The participants' liver disease history and associated person liver disease history data will be listed. Use of acetaminophen during the study, which has potential for hepatotoxicity, will be listed. Results from any hepatic monitoring procedures, such as a magnetic resonance elastography scan, and biopsy assessments will be listed, if performed.

Hepatic risk factor assessment data will be listed. Liver related signs and symptoms data will be summarized by treatment and listed. Alcohol and recreational drug use data will also be listed.

All hepatic chemistry, hematology, coagulation, and serology data will be listed. Values outside the reference ranges will be flagged on the individual participant data listings.

### 9.4.7 **Palatability Questionnaires**

The participant will be asked to provide responses to questions designed to assess the acceptability and palatability of the RTU suspension. The questionnaire will assess the participant's experience relating to the taste, smell, and after taste in the oral cavity.

The questionnaire will be completed by the participant immediately after administration of the RTU suspension and PFOS formulations.

These data will be summarized by treatment, and listed.

### 9.4.8 Other assessments

All other safety assessments not detailed in this section will be listed but not summarized or statistically analyzed.

### 9.4.9 Safety and Tolerability Statistical Methodology

No inferential statistical analyses are planned.

### 10. **INTERIM ANALYSES**

No interim statistical analyses are planned. If an unplanned interim analysis is deemed necessary for reasons other than a safety concern, the protocol and SAP must be amended.

### 11. CHANGES FROM THE PROTOCOL SPECIFIED STATISTICAL ANALYSES

There were no changes from the protocol specified statistical analyses.

Statistical Analysis Plan CONFIDENTIAL Labcorp Study: 8445329 Protocol Reference: J2G-MC-JZJU

# 12. REFERENCES

1. International Conference on Harmonization of Technical Requirements for Registration of Pharmaceuticals for Human Use, ICH Harmonized Tripartite Guideline, Statistical Principles for Clinical Trials (E9), 5 February 1998.

2. International Conference on Harmonization of Technical Requirements for Registration of Pharmaceuticals for Human Use, ICH Harmonized Tripartite Guideline, Structure and Content of Clinical Study Reports (E3), 30 November 1995.

# 13. DATA PRESENTATION

# 13.1 Derived Parameters

Individual derived parameters (e.g. PK parameters) and appropriate summary statistics will be reported to three significant figures. Observed concentration data, e.g. C<sub>max</sub>, should be reported as received. Observed time data, e.g. t<sub>max</sub>, should be reported as received. N and percentage values should be reported as whole numbers. Median values should be treated as an observed parameter and reported to the same number of decimal places as minimum and maximum values.

# 13.2 Missing Data

Missing data will not be displayed in listings.

# 13.3 Insufficient Data for Presentation

Some of the TFLs may not have sufficient numbers of participants or data for presentation. If this occurs, the blank TFL shell will be presented with a message printed in the center of the table, such as, "No serious adverse events occurred for this study."

Statistical Analysis Plan Labcorp Study: 8445329 Protocol Reference: J2G-MC-JZJU

### 14. **APPENDICES**

# **Appendix 1: Document History**

| Status and Version | Date of Change | Summary/Reason for Changes |
|--------------------|----------------|----------------------------|
| Final Version 1.0 | NA | NA; the first version. |

NA = not applicable

# Leo Document ID = a5a04ab0-7a10-4942-afd2-0fffd07bd491

Approver: PPD

Approval Date & Time: 05-Nov-2021 10:40:04 GMT

Signature meaning: Approved

Approver: PPD

Approval Date & Time: 08-Nov-2021 10:04:58 GMT

Signature meaning: Approved

Approver: PPD

Approval Date & Time: 08-Nov-2021 16:19:24 GMT

Signature meaning: Approved

Approver: PPD

Approval Date & Time: 09-Nov-2021 10:17:42 GMT

Signature meaning: Approved